CLINICAL TRIAL: NCT04180514
Title: Applying Pulse Wave Analysis to Predict Intradialytic Hypotension
Status: Completed | Type: Observational
Sponsor: China Medical University, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Han-Kuei Wu, Assistant Professor, School of Post-Baccalaureate Chinese Medicine, China Medical University, Taiwan
Other Study IDs: IDH-pulse
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Intradialytic Hypotension
Keywords: intradialytic hypotension; pulse wave analysis; heart rate variability; Constitution in Chinese Medicine Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intradialytic hypotension: subjects with intradialytic hypotension episode
  Interventions: Diagnostic Test: intradialytic hypotension episode
- Non-intradialytic hypotension: subjects without intradialytic hypotension episode

INTERVENTIONS:
Diagnostic Test: intradialytic hypotension episode — Intradialytic hypotension episode under regular hemodialysis
  Groups: Intradialytic hypotension

SUMMARY:
Intradialytic hypotension (IDH) is a common complication during hemodialysis in patients with chronic kidney disease and may increase the mortality. This study aimed to investigate whether pulse wave analysis could be the predictor of IDH.

In this study, patients under regular hemodialysis were enrolled from Taoyuan Chang Gung memorial hospital. Subjects were evaluated by pulse wave instrument, heart rate variability analyzer and Constitution in Chinese Medicine Questionnaire before hemodialysis. According to the definitions of IDH, subjects in study group and control group were confirmed by the dialysis records. Furthermore, repeated examinations were done for 3 hemodialysis to investigate the possible predictive factors for IDH.

DETAILED DESCRIPTION:
Intradialytic hypotension (IDH) is a common complication during hemodialysis in patients with chronic kidney disease and may increase the mortality. This study aimed to investigate whether pulse wave analysis could be the predictor of IDH.

In this study, patients under regular hemodialysis were enrolled from Taoyuan Chang Gung memorial hospital. Subjects were evaluated by pulse wave instrument, heart rate variability analyzer and Constitution in Chinese Medicine Questionnaire before hemodialysis. According to the definitions of IDH, subjects in study group and control group were confirmed by the dialysis records. Furthermore, repeated examinations were done for 3 hemodialysis to investigate the possible predictive factors for IDH.

ELIGIBILITY:
Inclusion Criteria:

* patients under regular hemodialysis (3 times per week) in last 3 months

Exclusion Criteria:

* arrhythmia
* artery-vein anastomoses on both arms
* other conditions which might interfere the evaluation of pulse wave analysis and heart rate variability analysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under regular hemodialysis in Chang Gung Memorial Hospital
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2016-12-17 (Actual)

PRIMARY OUTCOMES:
Pulse wave analysis | within 2 hours before regular dialysis
  Pulse wave analysis
Heart rate variability | within 2 hours before regular dialysis
  Heart rate variability
Constitution in Chinese Medicine Questionnaire | within 2 hours before regular dialysis
  Constitution in Chinese Medicine Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yang Chang, Doctor, Study Director — Chang Gung Memorial Hospital, Taoyuan, Taiwan.; Hen-Hong Chang, Doctor, Study Chair — China Medical University, Taichung; Han-Kuei Wu, Doctor, Principal Investigator — China Medical University, Taichung, Taiwan.; Hao-Min Cheng, Doctor, Study Director — Taipei Veterans General Hospital, Taipei, Taiwan.

IPD SHARING:
Plan to Share IPD: Undecided